CLINICAL TRIAL: NCT04453046
Title: Depleting Exosomes to Improve Response to Immune Therapy in Head and Neck Squamous Cell Cancer: An Early Feasibility Phase I Clinical Trial
Brief Title: Hemopurifier Plus Pembrolizumab in Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Eligible subjects at study site
Sponsor: Aethlon Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEMD-2019-01
Record Dates: First submitted 2020-06-20; First posted 2020-07-01 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Head- Neck Cancer; Hemopurifier; Pembrolizumab; Keytruda; Exosome; Immuno-oncology; Checkpoint inhibitor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This trial will evaluate the use of the Hemopurifier in combination with pembrolizumab (Keytruda) in patients with advanced and/or metastatic head and neck cancer. The Hemopurifier is a blood filtration device similar to a kidney dialysis cartridge which is designed to remove small particles called exosomes from the blood. Exosomes are believed to be involved in suppression of the immune system in cancer patients. The study will evaluate whether pretreatment with the Hemopurifier before administration of pembrolizumab is safe and well tolerated and results in lower numbers of exosomes in the blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Hemopurifier and Pembrolizumab (Experimental): In this clinical trial, the exosome-depleting device, the Hemopurifier, will be combined with standard of care therapy, Pembrolizumab. The purpose of the combination is to more effectively reduce immune suppression and provide a combined benefit of immune restoration for patients with recurrent/metastatic HNSCC. Therapy with the Hemopurifier will be initiated on the same day as and prior to Pembrolizumab infusion. The Hemopurifier treatment will be 4h. The subject treated with the Hemopurifier will remain in the Hemopurifier treatment area for the duration of the treatment. Pembrolizumab infusion will take place shortly after Hemopurifier treatment and may take place through the next day if needed.
  Interventions: Device: Hemopurifier; Drug: Pembrolizumab 200mg IV

INTERVENTIONS:
Device: Hemopurifier — Two Hemopurifier treatments on Day 1 and Day 21
Drug: Pembrolizumab 200mg IV — Pembrolizumab 200mg IV will be administered every 21 days. One cycle is 21 days. All patients will be treated with Pembrolizumab for up to 34 cycles

SUMMARY:
This is an Early Feasibility Study (EFS) investigating the use of the Hemopurifier to clear immunosuppressive exosomes in combination with pembrolizumab (Keytruda) in the front line setting, in patients with advanced and/or metastatic squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
All 12 patients enrolled into this Early Feasibility Phase I clinical trial will receive the same treatment of Hemopurifier plus Pembrolizumab (i.e., 2 rounds of Hemopurifier plus Pembrolizumab followed by Pembrolizumab only up to 2 years). Prior to initiation of the Hemopurifier treatment on Day 1, each subject will undergo phlebotomy to provide a baseline EDTA anti-coagulated blood sample, 30ml (< 3 tablespoons of blood) for the assessments of total exosome protein (TEP) levels and exosome profiles. The kinetics of exosome depletion will be evaluated in the study participants using serial blood samples (5ml) collected hourly during the 4h-depletion period by the Hemopurifier on Day 1. In addition, to evaluate kinetics of exosome recovery, 30ml of blood will be collected just prior to Pembrolizumab infusion (day 1) and on days 7 and 14 after Hemopurifier plus Pembrolizumab treatment during cycle 1 and 2. Exosome recovery after Hemopurifier + Pembrolizumab therapy will be evaluated and used to determine the rate of TEP recovery for each patient. Serial monitoring of TEP during Hemopurifier treatment (hourly during the 4h-depletion period), before Pembrolizumab infusion and after the second round of Pembrolizumab (days 7, and 14) will be done as for the first treatment. Only 2 Hemopurifier treatments will be given. For third and later rounds of Pembrolizumab, the investigators will continue to draw 30mL blood prior to Pembrolizumab infusion for the assessments of TEP levels and exosome profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent or metastatic HNSCC (oral cavity, oropharynx, larynx, hypopharynx) and not amenable to local therapy with curative intent (surgery or radiation therapy)
2. Qualifies for Pembrolizumab monotherapy as part of standard of care (has PD-L1 CPS ≥1)
3. ECOG performance status of 0-1
4. Measurable disease by RECIST 1.1
5. Be > 18 years of age on day of signing informed consent
6. Be willing and able to provide written informed consent for the trial
7. Life expectancy of at least 12 weeks based on investigator estimate
8. Adequate organ function as defined as:

   * WBC ≥ 2000/μL
   * Neutrophils ≥ 1500/μL
   * Platelets ≥ 100 x103/μL
   * Hemoglobin ≥ 8.0 g/dL
   * serum creatinine < 1.5 x ULN or creatinine clearance (CrCl) > 40 mL/min (using the Cockcroft-Gault formula)
   * AST/ALT < 3 x ULN
   * Total bilirubin < 1.5 x ULN (except subjects with Gilbert Syndrome who can have total bilirubin < 3mg/dL.
9. Women of childbearing potential (WCBP) must have a negative urine pregnancy test within 7 days prior to the first study intervention.
10. WCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and through 120 days after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for the duration of study participation.

    -

Exclusion Criteria:

1. Patients with salivary gland SCC or cutaneous SCC will be excluded
2. Has received systemic therapy (chemotherapy, immunotherapy, investigational therapy) for the treatment of recurrent/metastatic disease. Systemic therapy given concurrent with radiation treatment in the recurrent setting does not exclude the patient.
3. Untreated brain metastasis or leptomeningeal metastasis.
4. Tumor invades into the internal carotid artery or other major blood vessels whereby the treating investigator feels anti-coagulation is contraindicated.
5. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (Prednisone > 10mg or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
6. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic therapy or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
7. Has a history of non-infectious pneumonitis that required steroids, evidence of interstitial lung disease, or currently active non-infectious pneumonitis.
8. Has an active infection requiring systemic therapy.
9. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
10. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
11. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) in the recurrent/metastatic setting. Patients that received any of these agents in the upfront curative intent setting can be enrolled as long as it has been 1 year since the last dose.
12. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
13. Has known active Hepatitis B or active Hepatitis C
14. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
15. Concurrent therapy with an angiotensin-converting enzyme (ACE) inhibitor. ACE inhibitors must be discontinued at least 14 days prior to initiation of each Hemopurifier treatment and remain discontinued for 24 hours post treatment.
16. Systolic blood pressure less than 100 on at least 2 readings
17. Subjects with electro-cardiograms (ECG) showing clinically significant abnormalities.
18. Recent history of bleeding or bleeding disorders or any condition whereby in the opinion of the treating investigator giving anti-coagulation during the Hemopurifier treatment would be contraindicated
19. Any disorder or condition that in the opinion of the treating investigator would not be able to tolerate dialysis catheter placement, blood volume losses during Hemopurifier treatment or research blood draws.
20. History of heparin allergy or heparin induced thrombocytopenia.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Safety as measured by adverse events | Through study completion - Safety assessments will be completed at each study visits and up to two years after entry on protocol or until disease progression
  Safety will be determined in an Early Feasibility Phase I clinical trial for patients with recurrent/metastatic HNSCC who will undergo therapy with first line Pembrolizumab per standard of care combined with Hemopurifier treatments . All patients will be treated with Pembrolizumab every 21 days and, during active treatment, imaging will be done after every 3rd cycle as per standard of care. As part of the first two cycles of Pembrolizumab patients will receive Hemopurifier therapy immediately prior to Pembrolizumab infusion. The Hemopurifier therapy will last 4h and patients will receive their Pembrolizumab dose as soon as logistically possible, after Hemopurifier therapy on the same day.
Adverse Events | Day 1, Day 21, through study completion, up to two years
  Adverse events will be graded using CTCAE v5. The proportion of patients experiencing serious adverse events at least possibly related to treatment with Hemopurifier plus Pembrolizumab will be estimated with an exact 95% binomial confidence interval. Toxicity will be assessed continuously, and the trial will be paused if any patient experiences a treatment-related Grade 3 or worse adverse event. The rule is based on a beta-binomial model with an uninformative prior (α=1, β=1), where the trial is paused if P(P(Toxicity|Data and Prior)>0.3)>0.75.

SECONDARY OUTCOMES:
Levels of exosomes | Through study completion - up to two years after entry on protocol or until disease progression
  Kinetics of exosome depletion will be studied by drawing venous blood hourly starting immediately before, hourly during and immediately after each Hemopurifier treatment until Pembrolizumab treatment begins, for measuring total exosome protein level (TEP) and immunoinhibitory protein and miRNA profiles in the systemic circulation. Kinetics of exosome recovery will be studied by measuring TEP levels immediately prior to Pembrolizumab administration, and on days 7 and 14 after the first 2 cycles where patients are treated with Hemopurifier plus Pembrolizumab. Blood will be collected prior to each Hemopurifier treatment and each Pembrolizumab infusion for serial monitoring of TEP levels and immunoinhibitory protein and miRNA profiles.
Tumor response | Through study completion- up to two years or until disease progression
  CT imaging will be done after every 3rd cycle as per standard of car. If the patient 2 years of treatment and remains with CR/PR or SD, patient will undergo imaging every 3 months or sooner at the discretion of the treating physician. If a patient is taken off the study for progression, adverse events, or any other reason they will be seen 30 days afterwards for follow up followed by survival follow up every 3 months in the first year and every 6 months in the second year after withdrawal from study.
Survival | Through study completion - up to two years or until disease progression
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zandberg, MD, Principal Investigator — UPMC Hillman Cancer Center; Steven P. LaRosa, M.D., Study Director — Aethlon Medical Inc.
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No